CLINICAL TRIAL: NCT05030909
Title: An Integrated Transdiagnostic Protocol to Support Wellbeing in Adolescents From a Community Impacted by March 15 Attacks: a Randomized Controlled Trial
Brief Title: Feasibility Study of a Group Intervention for Youth Wellbeing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Collaborators: Canterbury Medical Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RO#21178
Record Dates: First submitted 2021-08-09; First posted 2021-09-01 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Psychological Distress; Trauma, Psychological; Emotional Problem
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Intervention Model Description: Trial Design This is a randomised control trial with a sequential waitlist control design to measure treatment effect sizes on primary and secondary outcomes of participant and parental wellbeing. We also will assess the methods of delivery, face validity and acceptability of treatment. Teenagers (aged 12-19) from the community will be recruited and allocated randomly to either two gender-specific groups to receive the same intervention over 6 weeks or to a comparison group who will be offered the intervention later. This balances the need for control groups while also widening access to the intervention for recruited participants. The study will be community-based in one site (Ōtautahi, Christchurch, New Zealand), with an emphasis on widening access to mental health supports in a minority community by maintaining cultural sensitivity and reducing stigma associated with mental illness.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transdiagnostic group protocol (Experimental): The study will run two gender-specific treatment groups (8 participants each) recruited from the community, with one individual session (for information, consent and initial data collection) and 6 group sessions. Both groups will receive the same intervention. A second round of recruitment will run later with anticipated n of 32 in the experimental arm.
  Interventions: Behavioral: transdiagnostic group treatment
- Waitlist control (Other): At both recruitment rounds, we will recruit 16 young people to receive the same intervention at a later stage. We will ask them to complete data collection at the same timepoints as the experimental arm participants to compare intervention effect size but will offer them the intervention afterwards so they still have access to the group. Data collected from them in the group will be used to assess feasibility and acceptability but not treatment effect size comparison.
  Interventions: Behavioral: transdiagnostic group treatment

INTERVENTIONS:
Behavioral: transdiagnostic group treatment — The individual and group sessions will integrate core principles from Motivational interviewing (provide information, address barriers), Cognitive Behavioural Therapy (psychoeducation regarding emotions, enhancing emotional awareness, cognitive restructuring, behavioural experiments, relaxation) , Acceptance Commitment Therapy (mindfulness, grounding, emotional and body awareness, enhancing cognitive flexibility), and aspects of Islamic psychology.

SUMMARY:
Psychological distress, anxiety and depression are common in adolescence, and even more so following traumatic events. On Friday 15 March 2019, two mosques in Ōtautahi, Christchurch were targeted in an act of terrorism, resulting in 71 people being injured and 51 people being shot dead. This has had widespread repercussions in the Muslim and wider community in Christchurch and New Zealand. Uptake of a response pathway set up by community and district health board groups has been low despite reports of high levels of distress in the adolescent population.

The proposed study offers a transdiagnostic group treatment approach (ie. Targeting a broad range of emotional difficulties) for teenagers from a community impacted by the March 15th shootings, incorporating well-evidenced transdiagnostic treatment principles into an Islamic Psychology framework to address the local population's need. We will determine the feasibility and effectiveness of this approach in increasing wellbeing in teenagers. We will run gender-specific treatment groups (8 participants in each group) recruited from the community, with one individual session (for information and consent) and 6 group sessions. We will measure symptoms of emotional difficulties, trauma symptoms and functioning at baseline, end of treatment and at 3 months follow-up. In addition, we will check in weekly with participants to monitor for any increased distress. We will also measure parental distress to explore whether an intervention for adolescents has an impact on parental wellbeing.

DETAILED DESCRIPTION:
Background and rationale On Friday 15 March 2019, two mosques in Christchurch were targeted in an act of terrorism. A white supremacist shooter attacked approximately 300 people, resulting in 51 deaths and 71 further people injured. The attack has been described as an attack on the Muslim faith and those affected by the event have expressed the importance of spiritual support as well as mental health support in the wake of the tragedy. Research into the effects of the attacks on adults in the Muslim community has identified significant concern over young people's mental health 1. A comprehensive framework of community support for children and adolescents was established involving collaboration between schools, primary care, community NGOs and secondary mental health services however the uptake of these services has been lower than expected despite reports of a growing need for support in these age groups1. Stigma regarding mental illness and distress has been identified as a major barrier to accessing supports.

Psychological distress, anxiety and depression are common in adolescence with substantial personal, societal and economic costs2,3. Transdiagnostic interventions (interventions which can be used across different mental health conditions) have gained support in treatment for adults, and evidence is emerging for their use in adolescent populations4-7. Evidence-informed holistic approaches to supporting wellbeing and mental health place less emphasis on pathology and can be more strengths-based with a focus on values. These approaches may appeal to young people and their families concerned about stigma and labelling 'difficulties' as 'disorders'.

Spiritually integrated psychotherapy has a growing evidence base and is associated with treatment adherence and therapeutic outcome8. An Islamic Psychology approach recognises spirituality as integral to the human experience, with models of Islamic psychotherapy gaining traction in recent years9. A model of traditionally integrated Islamic psychotherapy incorporates five interconnected elements; Áql (cognition), nafs (behavioural inclination), ruh (spirit), ihsas (emotion) and qalb (heart)10.

Holistic approaches to health are not new in New Zealand. Maori models of health are increasingly being adopted such as the Te Whare Tapa Wha model, emphasizing four cornerstones of Maori health11. These include Taha tinana (physical health), Taha wairua (spiritual health), Taha whanau (family health) and Taha hinengaro (mental health).

The proposed study offers a novel treatment approach for teenagers affected by the shootings, incorporating well-evidenced transdiagnostic treatment principles into an Islamic psychology framework to address the local population's need. It will assess the likely size of treatment effect on reported emotional difficulties and post-traumatic stress symptoms, and the feasibility of this approach in supporting wellbeing. We also will measure parental distress (mental health difficulties and physical symptoms) to explore whether an intervention for adolescents has an impact on parental wellbeing. The programme will also provide the opportunity to screen and identify individuals who may benefit from referral to further supports.

ELIGIBILITY:
Inclusion Criteria:

* All high school enrolled teenagers
* English speaking
* Participants do not need to identify as Muslim but will be made aware that the protocol incorporates elements of the Muslim faith.

Exclusion Criteria:

* active psychosis,
* severe substance use,
* intellectual disability
* non-English speaking young people.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — There will be two gender-specific groups. Participants will be able to choose which group they identify with (boy or girl). This is to increase acceptability within the Muslim culture.
Enrollment: 64 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Total problems score | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in total problems score in Strengths and Difficulties Questionnaire (SDQ), self report and parent report.Scored 0-40 with higher scores indicating more problems.
Emotional problems subscore | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in emotional problems subscore in Strengths and Difficulties Questionnaire (SDQ), self report and parent report. Score ranges 0-10 with higher scores indicating more emotional difficulties.
Trauma symptoms | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in total score of Child Revised Impact of Event Score (8 item ) (CRIES-8) by self report, score range 0-40, higher scores indicate more PTSD symptoms.
Somatic Symptom burden | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in somatic symptoms measured using Somatic Symptom Scale (8-item) (SSS-8) self report questionnaire by participants and parents. 5 point Likert scale gives a total score with range 0-32. Cutoff scores identify individuals with low (4-7), medium (8-11), high(12-15), and very high (16-32)somatic symptom burden.
Functional assessment | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in function measured using Children's Global Assessment Scale (CGAS) by clinician. Clinicians give a single global score ranging from 0-100 with higher scores indicating better functioning.
Time to recruitment | Measured before first group session at week 3.
  Time in weeks required to enrol 16 participants and hold initial individual session.
Implementation | Each session will be audio-recorded and scored (at individual session at week 1, weekly group sessions weeks 3- 7, and 3 month follow up/week 19)
  measured by use of fidelity scale to rate adherence to planned session content
Psychological flexibility | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in score on Acceptance and Action Questionnaire (AAQ-2), self
Awareness of experience | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in score on Awareness Indicator (AI), new measure asking about awareness of thoughts(aql), body sensations, feelings/emotions, and spiritual heart (qalb and ruh)

SECONDARY OUTCOMES:
Parental distress | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in distress measured using Kessler 10 (K-10) psychological questionnaire by parental self report and measured to identify whether further referrals are required. 5 point Likert scale gives a score of 10-50 with higher scores indicating higher distress. Scores 20-24 indicate likely mild mental disorder, 25-29 indicates likely moderate mental disorder and scores 30 and above indicate likely severe mental disorder. Referral will be offered for any scores over 20.
Suicidal risk | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  measured using Ask Suicide-screening questionnaire by self-report to assess whether further intervention is necessary and for any deterioration in mental state.It has 4 screening questions and a positive response to any of the 4 questions indicates a positive screen.
Participant Wellbeing | at each individual (week 1) and group session (weeks 3-7) and at 3 month follow up (week 19).
  measured using the Child Outcome Rating Scale (CORS) by self report to check for any deterioration in wellbeing. The CORS is a 4 item visual analogue scale to give a quantitative measure of individual wellbeing, relationships, social role and overall wellbeing.
Personality traits | three time points - initial individual session at week 1, final group session at 7 weeks and 3 month follow up (week 19).
  change in specific traits of Extroversion, Neuroticism, Openness, Conscientiousness Agreeableness measured using the Big Five Inventory - 10 item (BFI-10) measure by self report. 10 questions are answered on a 5 point Likert scale giving a score for each personality trait.
Attendance rates | recorded at each weekly group session (weeks 3-7) and data collection point (at individual session at week 1, final group session at 7 weeks and 3 month follow up/week 19).
  measured by recording attendance.
Participant experience/acceptability | After each individual (week 1) and weekly group session (weeks 3-7). A brief qualitative interview with each participant at the final group session at week 7 will also ask for their experience of the group.
  measured by Child Session Rating Scale (CSRS) which uses a 4 item visual analogue scale to give a quantitative measure of acceptability. Qualitative feedback will also be collected.
Retention | At final data collection point at week 19.
  measured by recording retention/drop-out rates.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Bell, MD, Study Director — University of Otago, Christchurch
Locations (1):
- Department of Psychological Medicine, University of Otago, Christchurch, Christchurch, Canterbury, New Zealand

IPD SHARING:
Plan to Share IPD: No